CLINICAL TRIAL: NCT02349880
Title: A Shared Decision-making Training for Inpatients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Johannes Hamann, PI, Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SDM-training
Record Dates: First submitted 2015-01-23; First posted 2015-01-29 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Schizophrenia; Schizo-affective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Active Comparator): 5 hour cognitive training
  Interventions: Behavioral: shared decision making training
- intervention (Experimental): 5 hour shared decision making training
  Interventions: Behavioral: shared decision making training

INTERVENTIONS:
Behavioral: shared decision making training

SUMMARY:
"Shared decision-making" is being promoted as a promising approach for engaging patients with schizophrenia in medical decisions and improving satisfaction and adherence.

To implement shared decision-making, both physicians and patients should commit to it and engage in a mutual decision process. Most research, however, has addressed interventions that either focus on the doctors' side (e.g. "communication skills") or on informing patients about treatment options (e.g. "decision aids"). These approaches have been shown to be feasible in clinical practice but had no strong effects on treatment patterns or adherence, possibly because they were insufficient to motivate and enable patients to engage actively in decision-making. Moreover, these interventions still rely on the doctor's willingness to share decisions, which has been shown to vary considerably.

To overcome these limitations and since many patients do not feel competent to participate in decision-making we developed an intervention that focuses on patients' communicative competencies. this intervention, a five session group-training, will be implemented for inpatients suffering from schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65
* icd diagnosis F2
* sufficient German language skills

Exclusion Criteria:

* debility

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
adherence to antipsychotic medication | 12 months